CLINICAL TRIAL: NCT02645006
Title: Effectiveness of an Intervention by a Health Education Workshop Compared With the Usual Advice to Reduce the Incidence of Falls in Independent 65 Years and Older Not Institutionalized. Primary Prevention.CHANGING TO NEVER FALL. CTNF
Brief Title: Workshop for Primary Prevention of Falls. CHANGING TO NEVER FALL. CTNF
Acronym: CTNF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sociedad Madrileña de Medicina de Familia y Comunitaria (Other)
Collaborators: Comunidad de Madrid (Other)
Responsible Party: Principal Investigator, MARIA MEDINA SAMPEDRO, Especialista en Medicina Familiar y Comunitaria, Máster en Investigación en Atención Primaria, Coordinadora del Grupo de trabajo de Atención al Mayor de Somamfyc, Sociedad Madrileña de Medicina de Familia y Comunitaria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SomamfycCTNF
Record Dates: First submitted 2015-12-29; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Dietary Habits; Accidental Falls; Unspecified Fall, Occurrence at Home; Physical Activity
Keywords: falls; elderly; Exercise,Physical; vitamin d; home hazards; mediterranean diet; body mass index; lower extremity exercise movement technics; vitamin D intake; Short Physical Performance Battery (SPPB o Test de Guralnik)
MeSH Terms: conditions — Feeding Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention arm- 3 session workshop (Experimental): The intervention group will attend a three session workshop, will learn to recognize their risk factors for fall, will be encouraged to adopt a healthy diet (vitamin D consumption), modify home hazards , and increase physical activity (a strength and balance program at home and a group walking route). After a monthly telephone follow-up they are invited to attend a recall session, were they realize the change in the strength and balance tests results.
  Interventions: Behavioral: 3 session workshop
- Control arm- 1 session workshop (Other): The control group will attend a single workshop session summarizing the major points of prevention of falls ( risk factors of fall, healthy diet and vitamin D consumption, home hazards, physical activity). After a monthly telephone follow-up they are invited to attend the three session workshop for further prevention
  Interventions: Behavioral: 1 session workshop

INTERVENTIONS:
Behavioral: 3 session workshop — The intervention group will attend a three session workshop, will learn to recognize their risk factors for fall, will be encouraged to adopt a healthy diet (vitamin D consumption), modify home hazards , and increase physical activity (a strength and balance program at home and a group walking route). After a monthly telephone follow-up they are invited to attend a recall session, were they realize the change in the strength and balance tests results.
  Arms: Intervention arm- 3 session workshop
Behavioral: 1 session workshop — The control group will attend a single workshop session summarizing the major points of prevention of falls ( risk factors of fall, healthy diet and vitamin D consumption, home hazards, physical activity). After a monthly telephone follow-up they are invited to attend the three session workshop for further prevention.
  Arms: Control arm- 1 session workshop

SUMMARY:
The purpose of this study is to determine whether a primary prevention workshop is effective decreasing at least 13% the annual incidence of falls in elderly compared to the habitual counseling.

Before the first fall incident, the elderly aged 65 or more, living in community, are invited to attend a workshop on fall preventing activities and factor risk detection. This activity consists on four sessions (one session per week during three weeks and the fourth session one year later) in which the elderly are expected to detect their own fall risk factors, encouraged to introduce healthy habits and to increase physical activity in order to improve strength and balance specifically.

This workshop has been prepared by family physicians following the latest scientific recommendations, it will be lead by them on the first edition, but it has not been written in formal language in order to be used by volunteers concerned about aging topics, independent from the Health Service.

DETAILED DESCRIPTION:
This study is a Clinical Trial. The methodology is to compare the incidence of falls in two groups. The intervention group will attend a three session workshop, will learn to recognize their risk factors for fall, will be encouraged to adopt a healthy diet (vitamin D consumption), modify home hazards , and increase physical activity (a strength and balance program at home and a group walking route). After a monthly telephone follow-up they are invited to attend a recall session, were they realize the change in the strength and balance tests results.

The control group will attend a single workshop session summarizing the major points of prevention of falls ( risk factors of fall, healthy diet and vitamin D consumption, home hazards, physical activity). After a monthly telephone follow-up they are invited to attend the three session workshop for further prevention.

GOALS

GENERAL Evaluate the effectiveness of an intervention program in the form of health education workshop to reduce the incidence of falls in independent population aged 65 and older living in the community.

SPECIFIC:

1. Estimate and compare the effectiveness of the intervention program in a workshop on health education from a simple intervention with respect to:

   • Final results: Principal: number and percentage of falls regular physical exercise 150 minutes a week of aerobic exercise and two times a week strength training.

   Improvement of body mass index. Contribution supplement or vitamin D. Improved test scores Short Physical Performance Battery (SPPB or test Guralnik)

   • Intermediate outcomes: Reduction in the number of risks identified in the home. assistance to physical exercise as a group. Maintenance or support group for physical exercise. Reduction of fear of falling (Fall Efficacy Scale abbreviate) Improved quality of life (EuroQol 5) attendees know how to get up after a fall.
2. Select volunteers in the audience who wish to train to develop new editions of the workshop as teachers, reaching the Community dimension of primary prevention, under the supervision of the research group.
3. Other:

   * Knowledge: Identify the general risk factors for falls. Identify personal risk factors for falling. Identify the drugs associated with increased risk of falls.
   * Attitudes: Guide in avoiding risk factors and circumstantial household falls. Recognize lifestyle that favor falls. Reinforce the practice of daily physical activity. Encourage changes towards a balanced diet. Reviewing the reasons for fear of falling. Support the creation of self-help groups that encourage physical exercise daily.
   * Skills: Apply the advice received in the housing and clothing. Demonstrate that you know develop a balanced and healthy menu daily. Demonstrate that you know off the ground after a fall.

METHODOLOGY

Experimental study types randomized clinical trial, controlled, parallel with simultaneous monitoring of both groups. The scope of the study is the community, the social network to which they belong major centers of the Community of Madrid Random assignment of senior centers where the intervention groups of intervention and control is performed.

Masking of participants on receiving the intervention is done, and there is masking the analysis of statistical data by ignoring what group they belong results. The selection criteria of the subjects are wide to allow extrapolation of results, increasing the external validity of the study.

The intervention is a three-session workshop that explores the detection and correction of risk factors for falls, changing working habits related to falls and applying interventions that have been shown to be effective in the literature. Working knowledge, attitudes and skills. It follows a period of one year follow up with monthly phone call to know the existence of falls in that period and a session assessing memory with changes. The intervention which is compared with the group counseling reporting the risk factors associated with falls and the necessary interventions on the habits associated with them. Working knowledge without delving into the changing attitudes. Follow up with the same frequency call is performed that intervention to publicize the existence of the group falls in that period.

In terms of population, the selection will be made according to criteria of inclusion and exclusion, but recruitment is voluntary type. The workshop will promote the community level where the senior center selected as the site is located and workshop point to the interested persons. The inclusion period covering the two weeks prior to the date set for the workshop until the day before included. demographics (age, sex, cultural and socioeconomic status), data related to falls (if you have had a fall or previously, current treatment with vitamin D, concomitant diseases, associates, toxic drugs), accessibility data will be collected (residence next to the workshop venue, existence of stairs at home, time availability to attend all sessions, physical limitations to attend regardless).

Person 65 years or older, habitual residence (more than nine months per year) in the coverage area of the senior center participants, independent ambulation by the field without help from another person, able to attend: inclusion criteria defined all sessions, acceptance of telephone follow-up, commitment to attend the final session, and given their informed consent to participate in the trial.

Institutionalized person, moderate or severe cognitive impairment of any etiology, blindness, total deafness, trouble reading, absolute contraindication for exercise or surgery in the previous 6 months: exclusion criteria are defined.

The study variables are the following, in addition to the previously referred to as demographic, related to falls or Accessibility:

Previous falls yes / no, Alcohol yes / no, grams of alcohol / week Group of neuroleptic drugs, benzodiazepines, other. Number of drugs. Number of barriers identified as checklist.

Corrected number of barriers. Reduce alcohol consumption, perform the homework, complete their daily findings, conducted prior to the workshop activity (type of activity, minutes, times a week), nutritional Journal: points. Weight, height, BMI, waist circumference. Fall Efficacy Scale abbreviate - points, apply the advice received during the three sessions (Diet- yes / no, Exercising-yes / no risk Home Improvement yes / no), the group is formed and go during the three weeks of the workshop but. Make exercise properly off the ground yes / no, number of attempts. Vit D treatment prior. Previous physical activity. Stairs at home. Technical assistance to walk. Limitations to physical activity. Active disease. 5D EuroQol quality of life: points. Health today points. Existence of hazards in home zones.

The assignment of participants in the control group or the intervention group may not be random by the type of intervention proposed, but senior centers will be randomized to receive the workshop with the sequence of intervention or monitoring sequence. It will be made, by an outside professional to the research team, a random sampling of the list of the 32 Centres for the Elderly in the Community of Madrid. As the intervention meets a priori criteria of benefit in primary prevention, control group will receive three intervention sessions of the workshop at the end of the follow-up period of 12 months.

The participant will ignore the existence of the two kinds of workshop, so that masking is achieved, however, not be possible to sign the informed consent prior to allocation to an intervention or another. As the researcher who teaches the workshop will be impossible masking since it will give the workshop in a sequence or another. It can be made in a double-blind follow-up period to perform the same telephone survey in both groups by a researcher other than educational workshop. Statistical analysis and evaluation of responses for statistical development outside the study will be conducted, reaching a triple blind.

As for the follow-up period, it is known that primary prevention to evaluate this time has to be very long. We have established a period of one year follow-up because it is the minimum referred to in the literature to detect impact on reducing falls interventions regarding physical activity and intake of vitamin D. However the aim of the researchers is to extend monitoring phone in a second phase to complete the second year. Protocol ensures in a pattern of telephone calls and data collected identical in both groups, scoring the reason for stopping monitoring whenever possible.

The strategy of data analysis will take into account the exclusion of participants (such as physical limitations) and causes of abandonment or follow-up workshop. An analysis was done by intention to treat the participant maintaining the data in the group assigned regardless of the end of the workshop or not.

The calculated sample size is 316 participants, 158 participants in each arm. Comparison of two proportions, unilateral test (the intervention is superior to standard treatment), 95% confidence level, 80% statistical power, P1 (ratio -. Incidence of falls in the gr control or usual care) 25%, P2 (expected incidence of falls in the intervention group) 12% (13% reduction). Sample size (n) = 109, expected loss ratio 20%.

Design effect (30 subjects per center. ICC 0.05). Design effect = 1+ (30.01) * 0.05 = about 1.15. Design effect 109 * 1.15 = 126. Adding 20% of losses = 158 participants per arm.

This study is designed as a pragmatic trial, evaluated the effectiveness of the workshop for primary prevention of falls, with broad selection criteria and heterogeneous population, as the reality that is to be applied, favoring the generalization of the results.

As for the limitations provided for the study, one of which is the participation of healthy individuals, and in the prevention field that requires a greater number of participants, a longer follow-up and possible higher rate of default. Furthermore you risk to specific bias as participation. You may only select those people who come to senior centers and premises where cartels are exposed invitation, which will be a priori greatest assets and willing to activities and social relationships. It is planned around this limitation in later editions of the workshop, when the offer to other sensitized social partners on this issue expands.

Another limitation is the supply of vitamin D, which has proven effective in those who present higher deficits of this vitamin. However since it is an external study the health system will not be available prior analytical determination, or it may decide to supplement in 600 or 800 units a day but will opt to increase the level of contribution to the diet. However, to have a letter to the family physician Participant is expected that a percentage of the participants are evaluated for vitamin deficiencies or receive supplements of vitamin D. These data will be recorded to be taken into account in the analysis phase.

ELIGIBILITY:
Inclusion Criteria:

* person 65 years or older
* habitual residence (more than nine months per year) in the coverage area of the senior center participants,
* walk independently without help from another person,
* able to attend all sessions,
* acceptance telephone follow-up,
* commitment to attend the final session,
* and given their informed consent to participate in the trial.

Exclusion Criteria:

* institutionalized person,
* moderate or severe cognitive impairment of any etiology,
* blindness,
* total deafness,
* trouble reading,
* absolute contraindication for exercise or surgery in the previous 6 months,
* engaged in other activities such muscle strengthening or tai chi balance.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
% incidence of falls in a year | one year
  % of incidence of falls in a year

SECONDARY OUTCOMES:
score in Short Physical Performance Battery (SPPB o Test de Guralnik) | one year
dietary vitamin D intake | one year
score in Mediterranean diet adherence test SEEDO (Sociedad Española para el Estudio de la Obesidad) | one year
number of home hazards modification | one year
% body mass index BMI | one year
score FES-I test (Fall Efficacy Scale) | one year
Score short MNA_spanish (Mini Nutritional Assessment) | one year
Score EuroQol-5D (EQ-5D) | one year

CONTACTS AND LOCATIONS:
Overall Officials: María Medina-Sampedro, MD, Principal Investigator — Somamfyc, Sociedad Madrileña de Medicina Familiar y Comunitaria
Locations (1):
- Comunidad de Madrid, Centros de Mayores del SRBS, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568